CLINICAL TRIAL: NCT05202990
Title: Pilot Study of a New Technique of Oral Fecal Transplantation Using Frozen Stool Capsules for the Maintenance Treatment of Pediatric Ulcerative Colitis.
Brief Title: Oral Fecal Microbiota Transplantation in Pediatric Ulcerative Colitis
Acronym: T-FORE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: MRSU 938 - Research Center of Saint Antoine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180572; 2024-518044-20-00 (EU CTIS Number)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Ulcerative Colitis in Remission
Keywords: Ulcerative Colitis; Pediatric Onset Inflammatory Bowel Disease; Microbiota; Fecal Microbiota Transplantation; Stool capsule; Intra-rectal enemas
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal Microbiota Transplantation by Stool capsules (Experimental): Patients receiving fecal microbiota transplantation from a healthy donor in 3 times after inclusion and randomisation (Month 0 - Month 1 - Month 2) using frozen stool capsules
  Interventions: Drug: Fecal Microbiota Transplantation by Stool capsules
- Fecal Microbiota Transplantation by enema (Experimental): Patients receiving fecal microbiota transplantation from a healthy donor in 3 times after inclusion and randomisation (Month 0 - Month 1 - Month 2) using frozen stool enemas.
  Interventions: Drug: Fecal Microbiota Transplantation by Intra-rectal enemas

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation by Stool capsules — After colon cleansing using PolyEthylen glycol, the patient will have a colonoscopy under general anaesthesia.
  The patient will then receive orally FMT (frozen stools capsules prepared from healthy donor feces).
  Other Names: UC treatment
  Arms: Fecal Microbiota Transplantation by Stool capsules
Drug: Fecal Microbiota Transplantation by Intra-rectal enemas — After colon cleansing using Polyethylen glycol, the patient will have a colonoscopy under general anaesthesia.
  The patient will then receive first FMT (frozen preparation of stools) by infusion in caecum during colonoscopy and the second and third doses by enemas.
  Other Names: UC Treatment
  Arms: Fecal Microbiota Transplantation by enema

SUMMARY:
The purpose of this study is to evaluate whether FMT by frozen stool capsules in pediatric UC patients in remission after corticosteroid treatment, can modify their dysbiotic gut microbiota by increasing the richness of their microbiota at 6 months.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is characterized by chronic inflammation of the colon of undetermined origin. Their incidence is increasing dramatically in the paediatric population.

Pediatric-onset inflammatory bowel disease (IBD) is characterized by a greater severity than adult IBD. Although great progress has been made in recent years, the pathogenesis of IBD is not fully elucidated. During UC, an imbalance in the composition of gut microbiota, called "dysbiosis", has been identified. This dysbiosis is notably characterized by an increased proportion of pro-inflammatory microorganisms and a decreased proportion of anti-inflammatory microorganisms. The current treatments used in IBD mainly target the immune system through immunosuppressants, and help to shorten flairs and prevent recurrences, but there is no curative treatment.

From a therapeutic point of view, the correction of this dysbiosis is thus an attractive approach. Until now, efficacy of microbiome-based therapies such as probiotics or antibiotics has been disappointing in IBD. Fecal microbiota transplantation (FMT) consists of the administration of fecal material from a donor into the intestinal tract of a recipient to change their microbiota composition and restore healthy conditions. FMT has been successfully used for many years for the treatment of Clostridioides difficile infection. Recent studies seem to show a benefit of FMT in UC.

The investigator's main hypothesis is that the replacement of a dysbiotic microbiota by a 'healthy' microbiota by FMT can modify the richness of UC patient's microbiota and has a positive impact on the disease course.

Once steroid-induced remission will be achieved, patients will be included and randomised to receive either FMT by frozen stool capsules or enemas. They will receive 3 doses at 0, 1 and 2 months. They will be followed for one year with stool samples collected every 3 months. Clinical and laboratory data will be collected.

ELIGIBILITY:
Inclusion Criteria for patients:

* Patient aged 8 to 17 years old
* Ulcerative colitis (UC), whatever the extent, except isolated proctitis (<5 cm), diagnosed for more than 3 months according to the usual clinical, biological and endoscopic criteria
* Moderate active UC defined by a PUCAI score > 35 and responding to corticosteroid treatment with a PUCAI score <10 at enrollment
* Treatment of UC (5-ASA, immunosuppressants, biotherapies) stable for more than 3 months
* Patient able to swallow test capsules
* For girls of childbearing age:

  * To have a negative blood (or urine) pregnancy test
  * To agree to use a reliable contraceptive method from visit 1 until the end of the research
* Patient with health insurance
* Informed written consent form signed by both parents or by the person (s) with parental authority

Exclusion Criteria for patients:

* isolated proctitis (<5 cm)
* Being on enteral nutrition
* Have received antibiotic or antifungal treatment in the 4 weeks prior to enrollment
* Having a Clostridioides difficile infection in the 4 weeks prior to enrollment;
* Being pregnant or breastfeeding, or have a positive pregnancy test;
* Have a contraindication to colonoscopy or general anaesthesia

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Success of FMT with frozen stool capsules defined by an increase in the richness of the recipient's microbiota at 6 months. | 6 months after the first Fecal Microbiota Transplantation (FMT)
  Success of FMT is defined by an increase in the richness of the recipient's microbiota at 6 months. Microbiota richness will be evaluated by measuring the alpha diversity of the microbiota using Shannon index.
  The success of the FMT will be defined by an increase in the Shannon index of 0.5 points between the recipient microbiota at M0 and the recipient microbiota at M6.

SECONDARY OUTCOMES:
Success of FMT with frozen stool capsules defined by an increase in the richness of the recipient's microbiota at 12 months | 12 months after the first FMT
  The success of the FMT will be defined by an increase in the Shannon index of 0.5 points between the recipient microbiota at M0 and the recipient microbiota at M12.
Success of FMT by stool enema defined by an increase in the richness of the recipient's microbiota at 6 and 12 months | 6 and 12 months after the first FMT
  The success of the FMT will be defined by an increase in the Shannon index of 0.5 points between the recipient microbiota at M0 and the recipient microbiota at M6 and M12
Success of FMT with frozen stool capsules on the change of recipient dysbiotic microbiota at 6 and 12 months | 6 and 12 months after the first FMT
  The success of the FMT will be defined by a Bray Curtis (BC) Index [recipient after FMT vs donnor] greater than a BC Index [recipient after FMT vs recipient before FMT], with a BC Index [recipient after FMT vs donnor] ≥ 0.6.
Success of FMT by enema on the change of recipient dysbiotic microbiota at 6 and 12 months | 6 and 12 months after the first FMT
  The success of the FMT will be defined by a Bray Curtis (BC) Index [recipient after FMT vs donnor] greater than a BC Index [recipient after FMT vs recipient before FMT], with a BC Index [recipient after FMT vs donnor] ≥ 0.6.
Success of FMT with frozen stool capsules on the richness and change of mucosal microbiota at 12 months | 12 months
  The success of the FMT will be defined by an increase in the Shannon index of 0.5 points between the mucosal recipient microbiota at M0 and the mucosal recipient microbiota at M12
Success of FMT by enema on the richness and change of mucosal microbiota at 12 months | 12 months
  The success of the FMT will be defined by an increase in the Shannon index of 0.5 points between the mucosal recipient microbiota at M0 and the mucosal recipient microbiota at M12
Success of FMT with frozen stool capsules on the change of mucosal recipient dysbiotic microbiota at 6 and 12 months | 6 and 12 months after the first FMT
  The success of the FMT will be defined by a Bray Curtis (BC) Index [recipient after FMT vs donnor] greater than a BC Index [recipient after FMT vs recipient before FMT], with a BC Index [recipient after FMT vs donnor] ≥ 0.6.
Success of FMT by enema on the change of mucosal recipient dysbiotic microbiota at 6 and 12 months | 6 and 12 months after the first FMT
  The success of the FMT will be defined by a Bray Curtis Index [recipient after FMT vs donnor] greater than a BC Index [recipient after FMT vs recipient before FMT], with a BC Index [recipient after FMT vs donnor] ≥ 0.6.
FMT with frozen stool capsules Feasibility | At inclusion, 1 and 2 months after each FMT
  Number of capsules intake, facility of capsules intake, tolerance, intake duration
FMT by enema Feasibility | At inclusion, 1 and 2 months after each FMT
  Number of enemas, tolerance , enemas duration, difficulties related to the application of enemas
Ulcerative colitis clinical relapse | 6 and 12 months
  Defined as a Pediatric Ulcerative Colitis Activity Index (PUCAI) > 35, number of relapses during the follow-up, treatments received during the follow-up
Ulcerative colitis Endoscopic relapse | 12 months
  Defined as an Ulcerative Colitis Endoscopic Index of Severity (UCEIS) ≥ 2
Change of inflammatory blood markers from baseline to 12 months | At inclusion, 6, 9 and 12 months
  CRP, VS, Leucocytes levels
Change of faecal calprotectin from baseline to 12 months | At inclusion, 6, 9 and 12 months
  Calprotectin level
Change of patient's quality of life evaluated with IMPACT-3 questionnaire from inclusion until 12 months | At inclusion 2, 6, 9 and 12 months
  IMPACT-3 questionnaire of 35 closed questions - scale ranging from 1 to 5 for all answers - higher score suggesting better quality of life
Incidence of adverse events | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte PIGNEUR, MD, PhD, Principal Investigator — AP-HP - Department of Pediatric Gastroenterology Hepatology and Nutrition - Necker - Enfants Malades Hospital; Harry SOKOL, MD, PhD, Study Director — AP-HP, Department of Gastroenterology and Nutrition - Saint Antoine Hospital
Locations (3):
- France (3):
  - Department of gastroenterology, Armand Trousseau Hospital, Paris
  - Department of Pediatric Gastroenterology, Hepatology and Nutrition - Necker - Enfants Malades Hospital, Paris
  - Department of Pediatric Gastroenterology, Robert Debré Hospital, Paris

IPD SHARING:
Plan to Share IPD: No